CLINICAL TRIAL: NCT04812834
Title: Systematic Detection and Screening of the Frailty Degree in Patients Admitted to the Emergency Department Short Stay Unit
Brief Title: Screening of the Frailty Degree in the Emergency Department Short Stay Unit
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-FRA-2020-74
Record Dates: First submitted 2021-03-12; First posted 2021-03-24 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Frail Elderly Syndrome
Keywords: elderly; frailty; short stay unit
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Screen all those> 65 years of age admitted to the Short Stay Unit for frailty, and detect those who are potentially fragile.

DETAILED DESCRIPTION:
Demographic change has led to a change in the profile and age of hospitalized patients, an increase in age and in patients with multiple chronic diseases and more complex health needs is observed.

Frailty is known to impact patient health outcomes with medical and surgical procedures. Thus, frailty is correlated with a greater presence of delirium, longer stays, a greater requirement for complementary examinations, a greater presence of mortality and other post-surgical complications, more dependence, more risks derived from hospitalization, and a greater need for convalescence after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age admitted to the Short Stay Unit

Exclusion Criteria:

* Patients under 65 years of age admitted to the Short Stay Unit

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients admitted to the Short Stay Unit of a 550-bed Urban and University Tertiary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-02-24 (Estimated); Study Completion 2023-02-24 (Estimated)

PRIMARY OUTCOMES:
To know the degree of frailty with the frail VIG index in patients admitted to the short-stay unit | 12 months
  The Frail Vig index ("VIG" is the spanish/catalan abbreviation for Comprehensive Geriatric Assessment) is a new, more concise Frailty index for rapid geriatric assessment, which contains 22 simple questions that assess 25 different deficits. The Frail VIG index score assesses the degree of frailty as a continuous variable. The value of the Frail VIG index is between 0 (absence of frailty) and 0.7 (severe frailty)

CONTACTS AND LOCATIONS:
Overall Officials: Josep JA Montiel Dacosta, PhDs, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Searle SD, Rockwood K. What proportion of older adults in hospital are frail? Lancet. 2018 May 5;391(10132):1751-1752. doi: 10.1016/S0140-6736(18)30907-3. Epub 2018 Apr 26. No abstract available. PMID 29706363
- [Result] Amblas-Novellas J, Martori JC, Molist Brunet N, Oller R, Gomez-Batiste X, Espaulella Panicot J. [Frail-VIG index: Design and evaluation of a new frailty index based on the Comprehensive Geriatric Assessment]. Rev Esp Geriatr Gerontol. 2017 May-Jun;52(3):119-127. doi: 10.1016/j.regg.2016.09.003. Epub 2016 Oct 28. Spanish. PMID 28029467
- [Result] Amblas-Novellas J, Martori JC, Espaulella J, Oller R, Molist-Brunet N, Inzitari M, Romero-Ortuno R. Frail-VIG index: a concise frailty evaluation tool for rapid geriatric assessment. BMC Geriatr. 2018 Jan 26;18(1):29. doi: 10.1186/s12877-018-0718-2. PMID 29373968
- [Result] Chong E, Ho E, Baldevarona-Llego J, Chan M, Wu L, Tay L. Frailty and Risk of Adverse Outcomes in Hospitalized Older Adults: A Comparison of Different Frailty Measures. J Am Med Dir Assoc. 2017 Jul 1;18(7):638.e7-638.e11. doi: 10.1016/j.jamda.2017.04.011. Epub 2017 Jun 3. PMID 28587850
- [Result] Damluji AA, Forman DE, van Diepen S, Alexander KP, Page RL 2nd, Hummel SL, Menon V, Katz JN, Albert NM, Afilalo J, Cohen MG; American Heart Association Council on Clinical Cardiology and Council on Cardiovascular and Stroke Nursing. Older Adults in the Cardiac Intensive Care Unit: Factoring Geriatric Syndromes in the Management, Prognosis, and Process of Care: A Scientific Statement From the American Heart Association. Circulation. 2020 Jan 14;141(2):e6-e32. doi: 10.1161/CIR.0000000000000741. Epub 2019 Dec 9. PMID 31813278